CLINICAL TRIAL: NCT03332433
Title: High-flow Nasal Cannula Oxygenation Decrease Hypoxia in Gastroscopy Sedated by Propofol: a Randomized Multicentre Clinical Trial
Brief Title: High-flow Nasal Cannula Oxygenation Decrease Hypoxia in Gastroscopy Sedated by Propofol
Acronym: HONCHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Pudong New Area People's Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, diansan su, Vice Chair of the Department of Anesthesiology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RenJiH-20170724
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Hypoxia; Gastric Cancer; Esophagus Cancer; Adverse Event
Keywords: Hypoxia; Gastroscope; High-flow nasal cannula
MeSH Terms: conditions — Hypoxia; Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Oxygen(2L/min) supplied with nasal catheter
- High-flow nasal cannula group (Experimental): Oxygen(up to 60L/min) supplied with high-flow nasal cannula
  Interventions: Device: High-flow nasal cannula oxygenation

INTERVENTIONS:
Device: High-flow nasal cannula oxygenation — Oxygen is supplied with a high-flow nasal cannula oxygenation device，the flow is up to 60L/min
  Arms: High-flow nasal cannula group

SUMMARY:
Hypoxia is the most common adverse events during sedated gastroscopy. In present study, high-flow nasal cannula oxygenation will be utilized in order to reduce the hypoxia. At the same time the feasibility and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing gastroscope
* age over 18 years old
* Signed informed consent form

Exclusion Criteria:

* Coagulation disorders or a tendency of nose bleeding;
* An episode/exacerbation of congestive heart failure (CHF) that requires a change in medication, diet or hospitalization from any cause in the last 6 months;
* Severe aortic stenosis or mitral stenosis;
* Cardiac surgery involving thoracotomy (e.g., coronary artery bypass graft (CABG), valve replacement surgery) in the last 6 months;
* Acute myocardial infarction in the last 6 months;
* Acute arrhythmia (including any tachycardia - or bradycardia) with hemodynamic instability;
* Diagnosed chronic obstructive pulmonary disease or current other acute or chronic lung disease requiring supplemental chronic or intermittent oxygen therapy);
* Increased intracranial pressure;
* ASA >III;
* Mouth, nose, or throat infection;
* Fever, defined as core body temperature > 37.5oC ;
* Pregnancy, breastfeeding or positive pregnancy test
* Emergency procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2034 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  (75% ≤ SpO2 < 90% for <60 s)

SECONDARY OUTCOMES:
Incidence of subclinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  (90% ≤ SpO2 < 95%)
Incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  (SpO2 < 75% for any duration or 75% ≤ SpO2 < 90% for >/=60 s)
Other adverse events | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Other adverse events include other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force and HFNC supportive oxygen therapy-related adverse events.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Renji hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Lin Y, Zhang X, Li L, Wei M, Zhao B, Wang X, Pan Z, Tian J, Yu W, Su D. High-flow nasal cannula oxygen therapy and hypoxia during gastroscopy with propofol sedation: a randomized multicenter clinical trial. Gastrointest Endosc. 2019 Oct;90(4):591-601. doi: 10.1016/j.gie.2019.06.033. Epub 2019 Jul 3. PMID 31278907